CLINICAL TRIAL: NCT01523639
Title: A Randomized, Placebo-controlled, Double-blind Multicenter Phase II Study to Investigate the Protectivity and Efficacy of Metformin Against Steatosis in Combination With FOLFIRI and Cetuximab in Subjects With First-line Palliative Treated, KRAS-Wild-Type, Metastatic Colorectal Cancer
Brief Title: A Randomized, Placebo-controlled, Double-blind Phase II Study Evaluating if Glucophage Can Avoid Liver Injury Due to Chemotherapy Associated Steatosis
Acronym: G-LUCAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Prematurely due to slow recruitment (07/08/2013). Newly defined study end=LPLV=05/11/2013. ABCSG guaranteed completed treatment period for ethical reasons.
Sponsor: Austrian Breast & Colorectal Cancer Study Group (Network)
Collaborators: Merck Gesellschaft mbH, Austria (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: G-LUCAS; 200084-610 (Other: Merck); 2011-001010-34 (EudraCT Number)
Record Dates: First submitted 2012-01-26; First posted 2012-02-01 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer; Steatohepatitis
Keywords: liver injury; steatosis; KRAS-Wild-Type; metastatic colorectal cancer; metformin; placebo; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Fatty Liver | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): FOLFIRI + cetuximab + metformin every 2 weeks for 12 cycles
  Interventions: Drug: Metformin/Placebo
- Placebo (Placebo Comparator): FOLFIRI + cetuximab + placebo every 2 weeks for 12 cycles
  Interventions: Drug: Metformin/Placebo

INTERVENTIONS:
Drug: Metformin/Placebo — The starting dose of Metformin/Placebo is 500 mg p.o. twice daily for 7 days (daily dose 1000 mg p.o.). Dose will be increased to 1000 mg p.o. twice daily at day 8 (daily dose 2000 mg p.o.) unless no toxicity ≥ 2 due to IMP occurs.
  Duration of treatment: 24 weeks
  Other Names: Glucophage

SUMMARY:
This multicenter randomized, placebo-controlled phase II study will enroll 132 first-line palliative treated subjects with metastatic KRAS wild type CRC. Subjects with histologically confirmed, KRAS wild-type CRC without previous chemo-therapy for metastatic disease will be screened for this study.

Approximately 10 sites in Austria will participate in the study. Subjects will be randomized in a ratio of 1:1 into two groups.

DETAILED DESCRIPTION:
This multicenter randomized, placebo-controlled phase II study will enroll 132 first-line palliative treated subjects with metastatic KRAS wild type CRC.

Wild-type KRAS is required for study entry. Further target-related parameters, based on current scientific knowledge may be assessed.

Subjects are randomized to Arm A or Arm B Arm A: FOLFIRI in combination with cetuximab and metformin Arm B: FOLFIRI in combination with cetuximab and placebo

A liver biopsy of hepatic metastasis and normal liver tissue is planned before the first cycle and at the end of treatment; with regard to the primary study objective, these subjects are evaluable.

Both efficacy and safety data will be collected. The investigators will assess response to treatment every 8 weeks based on imaging.

Following permanent treatment cessation, subjects will be followed-up for survival.

One interim analysis for futility (54 evaluable patients) and in addition two safety analysis for evaluation of reported adverse events between the two treatment groups will be performed at two different timepoints (20 evaluable patients/54 evaluable patients).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female >= 18 years of age
* Diagnosis of histologically confirmed, KRAS "wild-type" adenocarcinoma of the colon or rectum
* Non-resectable metastatic colorectal carcinoma
* Either presence of at least one liver lesion measurable unidimensionally by CT scan or MRI or at least one resectable liver metastasis with non-resectable extrahepatic disease (as assessed within 3 weeks prior to randomisation)
* Subjects scheduled to receive cetuximab and FOLFIRI
* ECOG performance status of 0 - 1 at study entry
* Leukocytes >= 3.0 x 10^9/L and neutrophils >= 1.5 x 10^9/L, platelets >= 100 x 10^9/L, and hemoglobin >= 8 g/dL
* Bilirubin <= 1.5 x ULN
* ASAT and ALAT <= 5 x ULN

Exclusion Criteria:

* Brain metastasis (if suspected, brain scan indicated)
* Previous chemotherapy for the currently existing metastatic disease
* Known or newly diagnosed diabetes
* Patients with ACS within the last three months
* Stage 3 or 4 heart failure defined according to the NYHA criteria
* Uncontrolled angina
* Contraindications to metformin (renal impairment [eGFR <45 mL/min/1.73m^2], known hypersensitivity to metformin, acute illness [dehydration, severe infection, shock, acute cardiac failure]), and suspected tissue hypoxia
* Surgery (excl. diagnostic biopsy, central venous catheter) or irradiation within 2 weeks prior to study entry defined as given written informed consent
* Concurrent chronic systemic immune therapy, chemotherapy, or hormone therapy not indicated in the study protocol
* Administration of any investigational agent(s) within 4 weeks prior to study entry,
* Previous exposure to EGFR-pathway targeting therapy
* Acute or sub-acute intestinal occlusion or history of inflammatory bowel disease
* Known grade 3 or 4 allergic reaction to any of the components of the treatment
* Any concurrent malignancy other than non-melanoma skin cancer, or carcinoma in situ of the cervix. (Subjects with a previous malignancy but without evidence of disease for >= 5 years will be allowed to enter the trial)
* Pregnancy or lactation
* Inadequate contraception (male or female patients) if of childbearing or procreative potential
* Known drug abuse/ alcohol abuse
* Legal incapacity or limited contractual capacity Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2013-11 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Reduction in the chemotherapy-associated steatosis | up to 24 weeks
  Reduction in the chemotherapy-associated steatosis, as assessed by the steatosis subcore of NAFLD activity score (NAS)

SECONDARY OUTCOMES:
Progression Free Survival | up to 30 months
  PFS will be evaluated after final study visits. Subjects who terminate the study before their scheduled final study visits will be censored.
Overall Survival | up to 30 months
  OS will be evaluated after final study visits. Subjects who terminate the study before their scheduled final study visits will be censored.
Safety assessment of all randomized subjects with at least one administration of study treatment | up to 24 weeks
  All subjects who received at least one dose of IMP. Additional safety analyses of reported AEs will be performed after the evaluation of 20 and 54 patients (between the 2 treatment groups) at the time of interim analysis.
Occured Adverse Events of all randomized subjects with at least one administration of study treatment | up to 30 months
  All subjects who received at least one dose of IMP. Additional safety analyses of reported AEs will be performed after the evaluation of 20 and 54 patients (between the 2 treatment groups) at the time of interim analysis.
Objective response rate (CR/PR) | up to 24 weeks
  Objective response rate (CR/PR), as assessed by RECIST criteria, version 1.1
Reduction in chemo-therapy associated steatohepatitis (CASH) | up to 24 weeks
  Reduction in chemo-therapy associated steatohepatitis (CASH) as assessed by NAS

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Gruenberger, MD, Principal Investigator — Austrian Breast & Colorectal Cancer Study Group
Locations (7):
- Austria (7):
  - Medical University Graz, Oncology, Graz, Styria
  - Medical University Innsbruck, Internal Medicine, Innsbruck, Tyrol
  - Hospital St. Vinzenz, Zams, Tyrol
  - Hospital BHS Ried, Ried, Upper Austria
  - KH BHB Vienna, Vienna
  - Med. Univ. Vienna, General Hospital Vienna, Vienna
  - KH St. Josef KH, Vienna

REFERENCES:
- [Background] Colucci G, Maiello E, Leo S, Giuliani F, Pedicini A, Pezzella G, Valori V, Galetta D, Contillo A, Prete F. Biochemical modulation of fluorouracil with high dose methotrexate or folinic acid in advanced colorectal cancer patients. Gruppo Oncologico dell' Italia Meridionale (GOIM). Anticancer Res. 1994 Sep-Oct;14(5B):2157-62. PMID 7840516
- [Background] Saltz LB, Cox JV, Blanke C, Rosen LS, Fehrenbacher L, Moore MJ, Maroun JA, Ackland SP, Locker PK, Pirotta N, Elfring GL, Miller LL. Irinotecan plus fluorouracil and leucovorin for metastatic colorectal cancer. Irinotecan Study Group. N Engl J Med. 2000 Sep 28;343(13):905-14. doi: 10.1056/NEJM200009283431302. PMID 11006366
- [Background] Scheithauer W, Kornek GV, Raderer M, Schull B, Schmid K, Kovats E, Schneeweiss B, Lang F, Lenauer A, Depisch D. Randomized multicenter phase II trial of two different schedules of capecitabine plus oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2003 Apr 1;21(7):1307-12. doi: 10.1200/JCO.2003.09.016. PMID 12663719
- [Background] Douillard JY, Cunningham D, Roth AD, Navarro M, James RD, Karasek P, Jandik P, Iveson T, Carmichael J, Alakl M, Gruia G, Awad L, Rougier P. Irinotecan combined with fluorouracil compared with fluorouracil alone as first-line treatment for metastatic colorectal cancer: a multicentre randomised trial. Lancet. 2000 Mar 25;355(9209):1041-7. doi: 10.1016/s0140-6736(00)02034-1. PMID 10744089
- [Background] Giacchetti S, Perpoint B, Zidani R, Le Bail N, Faggiuolo R, Focan C, Chollet P, Llory JF, Letourneau Y, Coudert B, Bertheaut-Cvitkovic F, Larregain-Fournier D, Le Rol A, Walter S, Adam R, Misset JL, Levi F. Phase III multicenter randomized trial of oxaliplatin added to chronomodulated fluorouracil-leucovorin as first-line treatment of metastatic colorectal cancer. J Clin Oncol. 2000 Jan;18(1):136-47. doi: 10.1200/JCO.2000.18.1.136. PMID 10623704
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Van Cutsem E, Kohne CH, Hitre E, Zaluski J, Chang Chien CR, Makhson A, D'Haens G, Pinter T, Lim R, Bodoky G, Roh JK, Folprecht G, Ruff P, Stroh C, Tejpar S, Schlichting M, Nippgen J, Rougier P. Cetuximab and chemotherapy as initial treatment for metastatic colorectal cancer. N Engl J Med. 2009 Apr 2;360(14):1408-17. doi: 10.1056/NEJMoa0805019. PMID 19339720
- [Background] Adam R, Pascal G, Castaing D, Azoulay D, Delvart V, Paule B, Levi F, Bismuth H. Tumor progression while on chemotherapy: a contraindication to liver resection for multiple colorectal metastases? Ann Surg. 2004 Dec;240(6):1052-61; discussion 1061-4. doi: 10.1097/01.sla.0000145964.08365.01. PMID 15570210
- [Background] Abdalla EK, Barnett CC, Doherty D, Curley SA, Vauthey JN. Extended hepatectomy in patients with hepatobiliary malignancies with and without preoperative portal vein embolization. Arch Surg. 2002 Jun;137(6):675-80; discussion 680-1. doi: 10.1001/archsurg.137.6.675. PMID 12049538
- [Background] Jaeck D, Oussoultzoglou E, Rosso E, Greget M, Weber JC, Bachellier P. A two-stage hepatectomy procedure combined with portal vein embolization to achieve curative resection for initially unresectable multiple and bilobar colorectal liver metastases. Ann Surg. 2004 Dec;240(6):1037-49; discussion 1049-51. doi: 10.1097/01.sla.0000145965.86383.89. PMID 15570209
- [Background] Rubbia-Brandt L, Audard V, Sartoretti P, Roth AD, Brezault C, Le Charpentier M, Dousset B, Morel P, Soubrane O, Chaussade S, Mentha G, Terris B. Severe hepatic sinusoidal obstruction associated with oxaliplatin-based chemotherapy in patients with metastatic colorectal cancer. Ann Oncol. 2004 Mar;15(3):460-6. doi: 10.1093/annonc/mdh095. PMID 14998849
- [Background] Fernandez FG, Ritter J, Goodwin JW, Linehan DC, Hawkins WG, Strasberg SM. Effect of steatohepatitis associated with irinotecan or oxaliplatin pretreatment on resectability of hepatic colorectal metastases. J Am Coll Surg. 2005 Jun;200(6):845-53. doi: 10.1016/j.jamcollsurg.2005.01.024. PMID 15922194
- [Background] DeLeve LD, Shulman HM, McDonald GB. Toxic injury to hepatic sinusoids: sinusoidal obstruction syndrome (veno-occlusive disease). Semin Liver Dis. 2002 Feb;22(1):27-42. doi: 10.1055/s-2002-23204. PMID 11928077
- [Background] Zorzi D, Laurent A, Pawlik TM, Lauwers GY, Vauthey JN, Abdalla EK. Chemotherapy-associated hepatotoxicity and surgery for colorectal liver metastases. Br J Surg. 2007 Mar;94(3):274-86. doi: 10.1002/bjs.5719. PMID 17315288
- [Background] Moertel CG, Fleming TR, Macdonald JS, Haller DG, Laurie JA. Hepatic toxicity associated with fluorouracil plus levamisole adjuvant therapy. J Clin Oncol. 1993 Dec;11(12):2386-90. doi: 10.1200/JCO.1993.11.12.2386. PMID 8246027
- [Background] Parikh AA, Gentner B, Wu TT, Curley SA, Ellis LM, Vauthey JN. Perioperative complications in patients undergoing major liver resection with or without neoadjuvant chemotherapy. J Gastrointest Surg. 2003 Dec;7(8):1082-8. doi: 10.1016/j.gassur.2003.08.005. PMID 14675719
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Vauthey JN, Pawlik TM, Ribero D, Wu TT, Zorzi D, Hoff PM, Xiong HQ, Eng C, Lauwers GY, Mino-Kenudson M, Risio M, Muratore A, Capussotti L, Curley SA, Abdalla EK. Chemotherapy regimen predicts steatohepatitis and an increase in 90-day mortality after surgery for hepatic colorectal metastases. J Clin Oncol. 2006 May 1;24(13):2065-72. doi: 10.1200/JCO.2005.05.3074. PMID 16648507
- [Background] Masi G, Loupakis F, Pollina L, Vasile E, Cupini S, Ricci S, Brunetti IM, Ferraldeschi R, Naso G, Filipponi F, Pietrabissa A, Goletti O, Baldi G, Fornaro L, Andreuccetti M, Falcone A. Long-term outcome of initially unresectable metastatic colorectal cancer patients treated with 5-fluorouracil/leucovorin, oxaliplatin, and irinotecan (FOLFOXIRI) followed by radical surgery of metastases. Ann Surg. 2009 Mar;249(3):420-5. doi: 10.1097/SLA.0b013e31819a0486. PMID 19247029
- [Background] Sasaki M, Itatsu K, Minato H, Takamura H, Ohta T, Nakanuma Y. Flare-up of nonalcoholic steatohepatitis after hepatectomy resulted in hepatic failure in a patient with type 2 diabetes mellitus. Dig Dis Sci. 2007 Dec;52(12):3473-6. doi: 10.1007/s10620-006-9662-7. Epub 2007 Apr 3. No abstract available. PMID 17404845
- [Background] Neuschwander-Tetri BA, Caldwell SH. Nonalcoholic steatohepatitis: summary of an AASLD Single Topic Conference. Hepatology. 2003 May;37(5):1202-19. doi: 10.1053/jhep.2003.50193. PMID 12717402
- [Background] Adams LA, Lymp JF, St Sauver J, Sanderson SO, Lindor KD, Feldstein A, Angulo P. The natural history of nonalcoholic fatty liver disease: a population-based cohort study. Gastroenterology. 2005 Jul;129(1):113-21. doi: 10.1053/j.gastro.2005.04.014. PMID 16012941
- [Background] Bugianesi E, Leone N, Vanni E, Marchesini G, Brunello F, Carucci P, Musso A, De Paolis P, Capussotti L, Salizzoni M, Rizzetto M. Expanding the natural history of nonalcoholic steatohepatitis: from cryptogenic cirrhosis to hepatocellular carcinoma. Gastroenterology. 2002 Jul;123(1):134-40. doi: 10.1053/gast.2002.34168. PMID 12105842
- [Background] Pessaux P, Panaro F, Casnedi S, Zeca I, Marzano E, Bachellier P, Jaeck D, Chenard MP. Targeted molecular therapies (cetuximab and bevacizumab) do not induce additional hepatotoxicity: preliminary results of a case-control study. Eur J Surg Oncol. 2010 Jun;36(6):575-82. doi: 10.1016/j.ejso.2010.04.010. Epub 2010 May 7. PMID 20452168
- [Background] Parkin DM, Pisani P, Ferlay J. Global cancer statistics. CA Cancer J Clin. 1999 Jan-Feb;49(1):33-64, 1. doi: 10.3322/canjclin.49.1.33. PMID 10200776
- [Background] Köhne CH, Van Cutsem E, Wils J, et al. Irinotecan improves the activity of the AIO regimen in metastatic colorectal cancer: Results of EORTC GI Group study 40986. Proc AmSocClinOncol 2003;22:Abstract 1018
- [Background] Tournigand C, Louvet C, Quinaux E et al. FOLFIRI followed by FOLFOX followed by FOLFIRI in metastatic colorectal cancer (MCRC): final results of a phase III study. Proc Am Soc Clin Oncol 2001;20:124a (Abstract 494)
- [Background] Tournigand C, Andre T, Achille E, Lledo G, Flesh M, Mery-Mignard D, Quinaux E, Couteau C, Buyse M, Ganem G, Landi B, Colin P, Louvet C, de Gramont A. FOLFIRI followed by FOLFOX6 or the reverse sequence in advanced colorectal cancer: a randomized GERCOR study. J Clin Oncol. 2004 Jan 15;22(2):229-37. doi: 10.1200/JCO.2004.05.113. Epub 2003 Dec 2. PMID 14657227
- [Background] de Gramont A, Figer A, Seymour M, Homerin M, Hmissi A, Cassidy J, Boni C, Cortes-Funes H, Cervantes A, Freyer G, Papamichael D, Le Bail N, Louvet C, Hendler D, de Braud F, Wilson C, Morvan F, Bonetti A. Leucovorin and fluorouracil with or without oxaliplatin as first-line treatment in advanced colorectal cancer. J Clin Oncol. 2000 Aug;18(16):2938-47. doi: 10.1200/JCO.2000.18.16.2938. PMID 10944126
- [Background] Eric Van Cutsem et al., Cetuximab plus FOLFIRI in the treatment of metastatic colorectal cancer - the influence of KRAS and BRAF biomarkers on outcome: Updated data from the CRYSTAL trial, ASCO GI 2010, Abstract # 281
- [Background] Zhou G, Myers R, Li Y, Chen Y, Shen X, Fenyk-Melody J, Wu M, Ventre J, Doebber T, Fujii N, Musi N, Hirshman MF, Goodyear LJ, Moller DE. Role of AMP-activated protein kinase in mechanism of metformin action. J Clin Invest. 2001 Oct;108(8):1167-74. doi: 10.1172/JCI13505. PMID 11602624
- [Background] Lin HZ, Yang SQ, Chuckaree C, Kuhajda F, Ronnet G, Diehl AM. Metformin reverses fatty liver disease in obese, leptin-deficient mice. Nat Med. 2000 Sep;6(9):998-1003. doi: 10.1038/79697. PMID 10973319
- [Background] Bugianesi E, Gentilcore E, Manini R, Natale S, Vanni E, Villanova N, David E, Rizzetto M, Marchesini G. A randomized controlled trial of metformin versus vitamin E or prescriptive diet in nonalcoholic fatty liver disease. Am J Gastroenterol. 2005 May;100(5):1082-90. doi: 10.1111/j.1572-0241.2005.41583.x. PMID 15842582
- [Background] Uygun A, Kadayifci A, Isik AT, Ozgurtas T, Deveci S, Tuzun A, Yesilova Z, Gulsen M, Dagalp K. Metformin in the treatment of patients with non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2004 Mar 1;19(5):537-44. doi: 10.1111/j.1365-2036.2004.01888.x. PMID 14987322
- [Background] Angelico F, Burattin M, Alessandri C, Del Ben M, Lirussi F. Drugs improving insulin resistance for non-alcoholic fatty liver disease and/or non-alcoholic steatohepatitis. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD005166. doi: 10.1002/14651858.CD005166.pub2. PMID 17253544
- [Background] Duseja A, Das A, Dhiman RK, Chawla YK, Thumburu KT, Bhadada S, Bhansali A. Metformin is effective in achieving biochemical response in patients with nonalcoholic fatty liver disease (NAFLD) not responding to lifestyle interventions. Ann Hepatol. 2007 Oct-Dec;6(4):222-6. PMID 18007551
- See also: Click here for more information about this study: open studies — http://www.abcsg.at